CLINICAL TRIAL: NCT04964960
Title: Phase II Investigation of Use of CNS Active Pembrolizumab and Chemotherapy for Asymptomatic Brain Metastasis From Non-small Cell Lung Cancer (NSCLC)
Brief Title: Pembro+Chemo in Brain Mets
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: John L. Villano, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, John L. Villano, MD, PhD, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21-NEURO-11
Record Dates: First submitted 2021-07-06; First posted 2021-07-16 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer; Lung Cancer Metastatic; Brain Cancer; Cancer
MeSH Terms: conditions — Lung Neoplasms; Brain Neoplasms; Neoplasms | interventions — pembrolizumab; Taxes; Paclitaxel; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab with standard of care chemotherapy treatment (Experimental): Patients will receive 200mg or 400mg of Pembrolizumab (standard of care dosing at the discretion of treating physician) over thirty minutes on day 1 every three or six weeks with standard of care chemotherapy treatment (carboplatin, pemetrexed, paclitaxel, nab-paclitaxel).
  Interventions: Drug: Pembrolizumab; Drug: Nab paclitaxel; Drug: Paclitaxel; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is an immunotherapy that can help fight certain cancers.
  Other Names: Keytruda
Drug: Nab paclitaxel — Nab-paclitaxel is a taxane derivative that is an albumin-bound paclitaxel nanoparticle formulation that promotes microtubule assembly.
Drug: Paclitaxel — Paclitaxel is a taxane derivative that promotes microtubule assembly by enhancing the action of tubulin dimers, stabilizing existing microtubules, and inhibiting their disassembly, interfering with the late G2 mitotic phase, and inhibiting cell replication.
Drug: Pemetrexed — Pemetrexed is an antifolate agent that disrupts folate-dependent metabolic processes essential for cell replication.
Drug: Carboplatin — Carboplatin is a platinum compound alkylating agent which covalently binds to DNA and interferes with the function of DNA by producing interstrand DNA cross-links.

SUMMARY:
The goal of this study is to evaluate whether providing Pembrolizumab prolongs survival and preserves quality of life while minimizing side effects for patients with NSCLC with untreated asymptomatic brain metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lunch cancer (NSLC) with untreated asymptomatic brain metastases
* NSLC lacks oncogenic driver mutations
* Absence of new onset neurological symptoms
* Presence of fewer than ten intracranial lesions
* Each lesion measures three centimeters or less
* Life expectancy of greater than three months
* Adequate organ and marrow function
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Presence of oncogenic driver mutations
* Measurable lesion located within 10mm of the optic chiasm or optic nerve, or within the brainstem
* Known leptomeningeal involvement.
* Midline shift
* Serious non-healing wound, ulcer or bone fracture
* Baseline inability to participate or complete neurocognitive testing
* Major surgical procedure (including craniotomy and open brain biopsy) or significant traumatic injury within 14 days prior to registration
* Receipt of a non-CNS minor surgical procedure (e.g. core biopsy or fine needle aspiration) within three days prior to registration
* History of allergic reactions attributed to monoclonal antibodies (mAb), compounds of similar chemical or biologic composition to Pembrolizumab
* Clinically significant cardiovascular disease
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Villano, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab with standard of care chemotherapy treatment
Started | 3
Completed | 1
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Did not complete cycles | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab with standard of care chemotherapy treatment
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate
Description: Intracranial benefit defined as stable disease, partial response, and complete response
Time Frame: 6 months (baseline to 6 months)
Population: Number of participants enrolled at 6 month timepoint
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab with standard of care chemotherapy treatment
Number analyzed (Participants) | 2
Participants
  Stable Disease | 0
  Complete Response | 2
  Partial Response | 0

2. Secondary Outcome: Number of Participants With Overall Survival at 12-month Post-enrollment
Description: Overall survival at 12-month post-enrollment
Time Frame: 12 months
Population: participants enrolled at 12 month timepoint
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab with standard of care chemotherapy treatment
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: Change in Extracranial Disease Control
Description: Extracranial disease control rate (systemic): includes stable disease, partial response, and complete response.
Time Frame: 12 months (6 months post-enrollment, 12 months post-enrollment)
Population: participants enrolled at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab with standard of care chemotherapy treatment
Number analyzed (Participants) | 1
Participants | 1

4. Secondary Outcome: Change in Patient-reported Cognitive Functioning - Functional Assessment of Cancer Therapy-Cognitive (FACT-Cog)
Description: The FACT-Cog questionnaire was developed to assess perceived cognitive function and impact on quality of life (QOL) in cancer patients. The level of perceived cognitive impairments is measured on a four-point Likert scale (4 = several times a day to 0 = never) FACT-Cog has been widely administered across clinical settings and validated across different cultures and languages. Subjects can complete it in 5 minutes. A higher score indicates a better quality of life/cognitive function.
Time Frame: 12 months (Baseline and 12 months post enrollment)
Population: participant declined to complete the questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pembrolizumab with standard of care chemotherapy treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Quality of Life - Functional Assessment of Cancer Therapy-Brain (FACT-Br)
Description: The FACT-Br is a commonly used instrument measuring general quality of life (QOL) that reflects symptoms or problems associated with brain malignancies across 5 subscales. The level of well-being is measured on a four-point Likert scale (4 = very much to 0 = not at all). The measure yields information about total quality of life, as well as information about the dimensions of physical well-being, social/family well-being, emotional well-being, functional well-being, and disease-specific concerns. The score range is 0-200 where a higher score indicated a better quality of life. The FACT-Br is written at the 4th grade reading level, and subjects can complete it in 5-10 minutes.
Time Frame: 12 months (Baseline and 12 months post enrollment)
Population: participant declined to complete the questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pembrolizumab with standard of care chemotherapy treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Quality of Life - FACIT Fatigue Scale (FACIT-F)
Description: FACIT-F is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four-point Likert scale (4 = not at all fatigued to 0 = very much fatigued) with a score range of 0-52. Subjects can complete the questionnaire in 2-3 minutes and the higher the score, the better the quality of life.
Time Frame: 12 months (Baseline and 12 months post enrollment)
Population: participant declined to complete the questionnaire
Arm/Group | Pembrolizumab with standard of care chemotherapy treatment
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in Mild Cognitive Impairment (MoCA)
Description: Neurocognitive functioning will be evaluated utilizing the Montreal Cognitive Assessment (MoCA). MoCA assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Participants will complete the MoCA (estimated time 10 minutes). The MoCA is scored to obtain an item total, scores can range from 0 to 30 and score of 26 or above is considered normal.
Time Frame: 12 months (Baseline and 12 months post enrollment)
Population: participant declined to complete the questionnaire
Arm/Group | Pembrolizumab with standard of care chemotherapy treatment
Number analyzed (Participants) | 0

8. Secondary Outcome: Change in Performance Status
Description: Participant performance status will be evaluated utilizing the Eastern Cooperative Oncology Group (ECGO) performance status instrument. Performance status is graded from 0-5 where lower scores indicate better performance/patient daily living abilities.
Time Frame: 12 months (Baseline and 12 months post enrollment)
Population: participant declined to complete the questionnaire
Arm/Group | Pembrolizumab with standard of care chemotherapy treatment
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Immune Based Biomarker Activity
Description: PD-1 and several immune-based markers, such as cytotoxic T cells, will be measured and summarized descriptively. Correlations with PD-1 and between markers will be estimated using Pearson or Spearman's correlation coefficient. Exploratory association of these biological markers with DCR will be performed using two-group comparison tests. Adjustment for multiple testing due to several immune-based markers will be considered using Holm's p-value adjustment method.
Time Frame: 12 weeks (Baseline, 6 weeks after baseline, 6 weeks after prior collection)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Pembrolizumab with standard of care chemotherapy treatment
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab with standard of care chemotherapy treatment (N=3)
Atrial Fibrillation (Cardiac disorders) | 1
Cardiac disorders - Other (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Flu like symptoms (General disorders) | 1
Other (General disorders) | 1
Sinusitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Weight gain (Investigations) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Spasticity (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT04964960/Prot_SAP_000.pdf